CLINICAL TRIAL: NCT06191458
Title: Neonatal Exposure to Primaquine Through Breast Milk During Treatment in Postpartum Women
Brief Title: Postpartum Primaquine in Breast Milk
Acronym: PBC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAL23004
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2024-08

CONDITIONS: Postpartum Women
Keywords: Postpartum women; Primaquine; Pharmacokinetics; Healthy
MeSH Terms: interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primaquine (Experimental): Twelve healthy postpartum women who are breast feeding healthy neonates 48 hours - 5 days old will receive primaquine 0.5 mg/kg once daily for 14 days.
  Interventions: Drug: Primaquine

INTERVENTIONS:
Drug: Primaquine — Primaquine 0.5 mg/kg (Government Pharmaceutical Organization, Thailand) will be given once daily with food for 14 days. This is the dose recommended by the World Health Organization for radical cure of P. vivax in tropical regions. Doses will be directly supervised (DOT).

SUMMARY:
Plasmodium vivax and ovale infections both follow chronically relapsing courses, leading to cumulative morbidity and mortality. P. vivax is the second most common malaria worldwide, with an estimated 13.8 million cases annually, and there is increasing concern about severe illness and death in vulnerable populations.

Radical cure of P.vivax and P.ovale with 8-aminoquinolines is necessary to prevent relapse. The most widely 8-aminoquinoline is primaquine (7-14 day course), which has been used for almost 75 years. Its widespread use is hampered by the potentially severe haemolysis primaquine may trigger in individuals with glucose-6-phosphate dehydrogenase (G6PD) deficiency, the most common red blood cell enzyme deficiency in the world. Safe administration of primaquine requires at least 30% of normal G6PD activity to avoid significant hemolysis.

Screening for malaria is routine in pregnancy, leading to improved detection of P. vivax infections, but primaquine and is contraindicated in pregnancy. As a result, relapses of P. vivax are common in postpartum and lactating women. Normal G6PD activity levels in infants less than 6 months old have only recently been described and have only been established along the Thailand-Myanmar border. Most low-resource settings are therefore unable to determine infant G6PD status. Uncertainty about infant G6PD status means that breastfeeding women are rarely offered radical cure because of theoretical concerns about drug exposure through breast milk triggering haemolysis in breastfed infants and children with G6PD deficiency. Though neonates generally have higher G6PD activity than adults, increased haemolysis for a neonate could theoretically contribute to neonatal jaundice and anaemia.

Understanding drug exposure to a breastfeeding neonate is operationally important, as interventions that can be safely offered before women leave the hospital postpartum have higher uptake. Current World Health Organization guidelines advise against prescribing primaquine to lactating women if they are breastfeeding infants less than 6 months old, or breastfeeding infants with G6PD deficiency or unknown G6PD status.

DETAILED DESCRIPTION:
This is a prospective open-label, single site, dense pharmacokinetic study of primaquine (0.5 mg/kg daily for 14 days) taken by postpartum lactating women.

The study will take place the Shoklo Malaria Research Unit (SMRU), Mahidol Oxford Tropical Medicine Research Unit, Tak Province, Thailand. Pregnant women who access care at SMRU antenatal care will be invited to participate after delivery with their breastfed children. Recruitment will prioritize women with a history of P. vivax infection without radical cure, but will also accept healthy volunteers. All 12 lactating women and their breastfed neonates 48 hours - 5 days old will be G6PD phenotypically normal, confirmed by spectrophotometry.

Following informed consent, women attending SMRU antenatal care will be pre-screened during pregnancy for potential enrolment postpartum. Full screening must be repeated postpartum before enrolment.

Similar to the mothers, neonates will be pre-screened for eligibility using biosensor and Hb/Hct. Birth history will be reviewed to determine the absence of severe neonatal disease (neonatal sepsis, severe jaundice, significant birth asphyxia etc).

Mothers and neonates will be closely monitored for safety throughout the 28 day follow up period including regular assessments of adverse events, Hb, Hct and MetHb levels. If a neonate develops jaundice, treatment will follow the clinical guidelines of the site. The study sampling will continue as long as the baby is responding normally to phototherapy and inclusion in the study is not thought to interfere with clinical care. If methemoglobinemia is detected, it will be managed according to SMRU clinical protocol. Medication will be stopped if the participant is in the primaquine arm and a severe drug related AE occurs.

Pharmacokinetic (PK)sampling plan:

* Mothers: Dense PK venous blood and breast milk sampling will be performed during day 1 and 14; two blood samples and one breast milk sample will collected at a single timepoint on days 3, 5 and 8.
* Neonate: One capillary blood sample will be collected on the same days as maternal sampling.

PK drug measurements of primaquine, and carboxyprimaquine will be performed. Drug concentrations will be quantified by liquid chromatography coupled with tandem mass spectrometry (LC-MS/MS) using a validated assay according to regulatory guidelines.

This study is funded by Thrasher Research Fund, EW "Al" Thrasher award.

ELIGIBILITY:
Inclusion Criteria: Mothers

* Lactating woman >= 18 years old
* Planning to breastfeed for the duration of the study
* Breastfeeding one infant 48 hours - 5 days old
* Willingness and ability to comply with the study protocol for the duration of the study
* Can understand information about the study and provide consent

Inclusion Criteria: Infants

• Healthy neonate 48 hours - 5 days old

Exclusion Criteria: Mothers

* Known hypersensitivity to Primaquine (PMQ), defined as history of erythroderma/other severe cutaneous reaction, angioedema or anaphylaxis
* Known Glucose-6-phosphate-dehydrogenase (G6PD) deficiency in mother defined as G6PD activity <70% of normal male population median by spectrophotometry
* Presence of any condition which in the judgement of the investigator would place the participant at undue risk or interfere with the results of the study
* Screening Hct <33% by complete blood count (CBC)
* Known history of severe jaundice in a previous child
* Blood transfusion within the 3 months before screening

Exclusion Criteria: Infants

* Known Glucose-6-phosphate-dehydrogenase (G6PD) deficiency in neonate defined as G6PD activity <70% of normal male population median by spectrophotometry
* Presence of any condition which in the judgement of the investigator would place the participant at undue risk or interfere with the results of the study
* Screening Hct <40% by CBC
* Estimated gestational age at birth < 38 weeks
* Evidence of birth asphyxia (5 min Apgar score <7)
* Moderate or severe jaundice as defined as total serum bilirubin above treatment line on day 1 (before maternal dose)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy lactating woman aged more than or equal to 18 years old
Enrollment: 12 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-02-23 (Actual); Study Completion 2025-02-23 (Actual)

PRIMARY OUTCOMES:
Area under the time-concentration curve in milk | 14 days
  Area under the time-concentration curve (AUC) for primaquine in colostrum and transitional milk
Relative infant dose | 14 days
  Relative infant dose (RID) is a measure of the weight-adjusted dose of the study medication that the infant is exposed to via the breast milk. It is the most clinically relevant measure of the safety for a breastfed child of maternal medication use. RID for primaquine will be calculated using AUCs for drug in maternal plasma and colostrum, and transitional milk.

SECONDARY OUTCOMES:
Area under the time-concentration curve in plasma | 14 days
  Area under the time-concentration curve (AUC) of primaquine for mother and neonate (if measurable concentrations found in neonatal plasma).
Time to maximum concentration | 14 days
  Time to maximum concentration (Tmax) of primaquine for mother and neonate (if measurable concentrations found in neonatal plasma).
Peak plasma concentration | 14 days
  Peak plasma or maximum concentration reached (Cmax) of primaquine for mother and neonate (if measurable concentrations found in neonatal plasma).
Haematologic changes | 14 days
  Changes in haemoglobin (Hb), haematocrit (Hct) and methemoglobin (MetHb) in mothers and neonates over the period of drug exposure.
Number of adverse events | 14 days
  Number of adverse events (AEs) in mothers and neonates during the period of drug exposure.
Severity of adverse events | 14 days
  Severity of adverse events (AEs) in mothers and neonates during the period of drug exposure according to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Type of adverse events | 14 days
  Type of adverse events (AEs) in mothers and neonates during the period of drug exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Rose McGready, Ph.D, Principal Investigator — Shoklo Malaria Research Unit (SMRU)
Locations (1):
- Shoklo Malaria Research Unit (SMRU), Mae Ramat, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: Yes
All data will be published in the open access medical literature with the identity of the participants protected. Criteria for authorship will follow international guidelines. Following completion of the study, the database will belong to the PI and key co-investigators. The deidentified database, including individual participant data, may be made freely available to other researchers via the Oxford University Research Archive. The results of the study will be shared with the local community.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After completion of trial activities. PI will upload results within 12 months of the end of the trial declaration.
Access Criteria: SMRU and MORU Data Sharing Policies
URL: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing/moru-tropical-network-policy-on-sharing-data-and-other-outputs